CLINICAL TRIAL: NCT03835715
Title: Interventional, Open-label, Flexible-dose Study of Vortioxetine on Emotional Functioning in Patients With Major Depressive Disorder With Inadequate Response to SSRI/SNRI Treatment
Brief Title: Study With Vortioxetine on Emotional Functioning in Patients With Depression
Acronym: COMPLETE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17797A
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vortioxetine (Experimental)
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Flexible doses (10-20 mg) of vortioxetine; 10 mg during the first week which may be increased up to 20 mg week 2-8
  Other Names: Brintellix ®

SUMMARY:
The study will evaluate effectiveness of flexible dose vortioxetine 10-20 mg/day on emotional functioning in patients with MDD with an inadequate response to SSRIs/SNRIs.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a primary diagnosis of single or recurrent MDD according to DSM-5®. The current major depressive episode (MDE) must be confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has had the current MDE for <12 months.
* The patient has a Montgomery and Åsberg Depression Rating Scale (MADRS) total score ≥ 22 and ≤ 28 at the Baseline Visit.
* The patient has been treated with SSRI/SNRI monotherapy (citalopram, escitalopram, paroxetine, duloxetine or venlafaxine) for at least 6 weeks at adequate dose for the current MDE and with an inadequate response and is a candidate for a switch in the investigator's opinion.
* The patient wants to switch antidepressant treatment.
* The patient has an ODQ total score ≥50 at baseline, while on SSRI/SNRI monotherapy (prior to switch).
* The patient answered "Yes "to the screening question on emotional effects.

Exclusion Criteria:

- The patient has a significant risk of suicide according to the investigator's clinical judgment or has made an actual suicide attempt in the previous 6 months prior to Baseline

Other in- and exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 8 in Oxford Depression Questionnaire (ODQ) total score | From baseline to Week 8
  The ODQ is a patient-centred, self-report measure of emotional symptoms present in patients treated with antidepressants. The ODQ is a 26-item patient self-complete measure, spread over 3 sections and covering 5 dimensions of: not caring (NC), emotional detachment (ED), positive reduction (PR), general reduction (GR), and antidepressant as cause (AC). Response options are based on 5-point Likert scale with a score applied to each response.

SECONDARY OUTCOMES:
Change from baseline to Week 8 in MEI total score. | From baseline to Week 8
  The Motivation and Energy Inventory (MEI) is a 27-item scale initially developed and validated for the purpose of evaluating interventions to improve motivation and energy in patients with depression. The MEI assesses three domains: mental or cognitive energy, social motivation, and physical energy. Scoring Respondents use scales ranging from 0 (indicating that the behavior is never present) to 5 or 6 (a behavior or feeling that is present very frequently or all of the time). Items 3-11, 13-15, 17, and 18 are reverse-scored in order to ensure that higher scores indicate greater levels of motivation and energy. All items use either a 5- or 7-point Likert type response scale.
Change from baseline to Week 8 in DSST total score | From baseline to Week 8
  The Digit-Symbol Substitution Test (DSST) is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making and motor skills. The DSST is sensitive to cognitive impairments affecting attention, processing speed, and executive function (including working memory). The DSST consists of 133 digits and requires the subject to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted. The total score is the number of correct symbols and the total score ranges from 0 (less than normal functioning) to 133 (greater than normal functioning).
Change from baseline to Week 8 in ODQ domain scores (NC, ED, PR, GR, and AC) | From baseline to Week 8
  The Oxford Depression Questionnaire (ODQ) is a patient-centred, self-report measure of emotional symptoms present in patients treated with antidepressants. The ODQ is a 26-item patient self-complete measure, spread over 3 sections and covering 5 dimensions of: not caring (NC), emotional detachment (ED), positive reduction (PR), general reduction (GR), and antidepressant as cause (AC). Response options are based on 5-point Likert scale with a score applied to each response.
Change from baseline to Week 8 in MADRS total score | From baseline to Week 8
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome.
Change from baseline to Week 8 in SDS individual item scores (family, work, and social life) | From baseline to Week 8
  Sheehan Disability Scale (SDS) measures disability. Total scores are computed by summing scores from all 3 items. Total score ranges from 0 to 30, with higher scores indicating greater disability. Reduction in SDS scores therefore indicates better outcome.
Change from baseline to Week 8 in SDS total scores | From baseline to Week 8
  Sheehan Disability Scale (SDS) measures disability. Total scores are computed by summing scores from all 3 items. Total score ranges from 0 to 30, with higher scores indicating greater disability. Reduction in SDS scores therefore indicates better outcome.
Change from baseline to Week 8 in CGI-S score | From baseline to Week 8
  The Clinical Global Impression severity of illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
CGI-I score at Week 8 | at Week 8
  The Clinical Global Impression - global improvement CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement is drug-related or not.

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (23):
- France (7):
  - Office of Dr. Patrick Bourgoin (FR0011), Angoulême
  - Cabinet Psyche (FR0012), Douai
  - Centre Medical Ambroise Pare (FR0007), Élancourt
  - Dr. David Modavi Md, Office Of (FR0001), Toulouse
  - Private Practice Dr. Paule Khalifa (FR0010), Toulouse
  - GHS De Nancy - CPN Laxou (FR0006), Vandœuvre-lès-Nancy
  - Dr Karim Boutayeb MD, Office of (FR0009), Viersat
- Italy (3):
  - DSM Giulianova c/o ospedale di Giulianova (IT0004), Giulianova
  - Dipartimento Salute Mentale ASL Lecce (IT0006), Lecce
  - Universita degli Studi di Roma La Sapienza - Azienda Ospedaliera Sant Andrea (IT0013), Rome
- Lithuania (6):
  - JSC Romuvos Klinika (LT0002), Kaunas
  - Mental Health Centre Kaunas Outpatient Clinic (LT0005), Kaunas
  - JSC Nefridos klinika (LT0006), Klaipėda
  - Jsc Silutes Mental Health And Psychotherapy Center (LT0001), Šilutė
  - Antakalnis Psychiatric Consultation Centre (LT0003), Vilnius
  - PI Mental Health Center of Zirmunai (LT0004), Vilnius
- Spain (7):
  - Hospital Universitario Fundacion Alcorcon (ES0009), Alcorcón
  - Instituto Internacional de Neurociencias Aplicadas (ES0004), Barcelona
  - Centro De Salud Mental De Foios (ES0002), Foios
  - University of Oviedo (ES0011), Oviedo
  - Francesca Canellas Dols (ES0005), Palma de Mallorca
  - Hospital Clínico Universiatrio de Salamanca (ES0001), Salamanca
  - Centro De Especialidades A Doblada (ES0006), Vigo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christensen MC, Adair M, Loft H, McIntyre RS. The Motivation and Energy Inventory (MEI): Analysis of the clinically relevant response threshold in patients with major depressive disorder and emotional blunting using data from the COMPLETE study. J Affect Disord. 2023 Feb 15;323:547-553. doi: 10.1016/j.jad.2022.11.033. Epub 2022 Nov 14. PMID 36395989
- [Derived] Christensen MC, Fagiolini A, Florea I, Loft H, Cuomo A, Goodwin GM. Validation of the Oxford Depression Questionnaire: Sensitivity to change, minimal clinically important difference, and response threshold for the assessment of emotional blunting. J Affect Disord. 2021 Nov 1;294:924-931. doi: 10.1016/j.jad.2021.07.099. Epub 2021 Jul 31. PMID 34378539